CLINICAL TRIAL: NCT01018160
Title: Practice and Patient Compliance on the PPI(Proton Pump Inhibitors) Treatment of Gastroesophageal Reflux in South Korea: A Prospective Observational Study
Brief Title: Practice and Patient Compliance on the PPI (Proton Pump Inhibitors) Treatment of Gastroesophageal Reflux in South Korea
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015436
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Rabeprazole sodium; Gastroesophageal Reflux; GERD; Observational
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: Rabeprazole Sodium

INTERVENTIONS:
Drug: Rabeprazole Sodium — 10mg - 20mg tablet once or twice daily for 12 weeks

SUMMARY:
The purpose of this study is to examine the treatment profile of approximately 1,000 adult patients with gastroesophageal reflux who begin raberpazole sodium treatment for 4 months, and assess patients' adherence to the study drug.

DETAILED DESCRIPTION:
This study is a multicenter, open-labeled, prospective, phase IV, observational study for patients visiting the gastroenterology department. The purpose of this study is to examine the treatment profile of approximately 1,000 adult patients with gastroesophageal reflux (GERD) who begin raberpazole sodium treatment for 4 months and assess patients' adherence to the study drug. The primary objective is to examine the treatment profile of gastroesophageal reflux in the secondary or tertiary clinical center. The secondary objective is to examine GERD patients' adherence to the study drug (rabeprazole sodium) during the treatment period. Of the patients who visit the study centers and complain about gastroesophageal reflux symptoms during the study period, those who are deemed to need rabeprazole sodium administration at the investigator's discretion will be considered for this study. The main outcome measures are the patterns of gastroesophageal reflux management (eg. treatment duration of initial therapy etc) and the compliance of proton pump inhibitor treatment.The compliance data (number of tablets taken) will be calculated at the clinical visit by counting the number of dispensed tablets that are remaining. Also, investigators will observe the gastroesophageal reflux symptom free rate at the end of initial therapy, gastrointestinal (GI) symptom relief and safety information at each visit. Study period is up to 4 months. During the study, no standardized treatment is stipulated, and patients may receive any treatment considered by their physicians. Rabeprazole sodium 10 mg - 20 mg tablet once daily for 4months.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining about heartburn or acid regurgitation, the typical GERD symptoms, more than once a week
* After a full explanation about the observational study, patients who fully understand it and sign a written consent form

Exclusion Criteria:

* Patients who took rabeprazole sodium within the last four weeks
* Patients who are hypersensitive to the active ingredient of rabeprazole sodium or benzimidazole
* Patient with other digestive tract diseases other than GERD (gastrointestinal cancer, liver disease, pancreatic disease, peptic ulcer, inflammatory digestive tract diseases [in case of ulcer, however, scars from healed ulcer may be included])
* Patients with other severe accompanying diseases including renal impairment, cerebrovascular disease, cardiovascular disease and severe respiratory disease
* Patients who must constantly take Proton Pump Inhibitors other than rabeprazole sodium during study period
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the patients who visit the department of gastroenterology with gastroesophageal reflux disease and who need rabeprazole treatment according to the doctor's discretion
Sampling Method: Non-Probability Sample
Enrollment: 1197 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
GERD Symptom improvement | 4 weeks, 16 weeks

SECONDARY OUTCOMES:
Actual administrating dosage of PPI during the GERD treatment period | 16 weeks
Visit interval during the GERD treatment | 16 week
Duration of GERD initial therapy | 16 week
Ratio of GERD patients who received endoscopy | 16 week
Ratio of GERD patients who received PH Monitoring Test | 16 week

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.